CLINICAL TRIAL: NCT04649125
Title: Advanced Techniques For Single-fraction Palliative Radiotherapy Versus Standard Multi Fraction Radiation
Acronym: ASPIRE_Multi
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Royal North Shore Hospital (Other)
Collaborators: Northern Sydney and Central Coast Area Health Service (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ASPIRE Multi
Record Dates: First submitted 2020-11-24; First posted 2020-12-02 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Palliative Radiotherapy

STUDY DESIGN:
Intervention Model Description: Non Comparative Randomised Trial Randomised between standard dose multifractions (5-10#) and single fraction dose escalated palliative radiation therapy
Who Masked: Investigator
Masking Description: Investigators do not know which arm patients have been randomised to
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- standard (Active Comparator): standard radiotherapy 5 fractions
  Interventions: Radiation: dose escalation
- single fraction dose escalation (Experimental): 8Gy to Planned Target Volume, 12Gy to Clinical Target Volume +/- 14Gy to Gross Target Volume
  Interventions: Radiation: dose escalation

INTERVENTIONS:
Radiation: dose escalation — single fraction dose escalation to the tumour

SUMMARY:
The aim of the study is to determine if single fraction dose escalated palliative radiotherapy results in a prolonged duration of benefit for patients otherwise suitable for Multifraction (5-10#) palliative radiation. The primary endpointis to determine the percentage of patients who have achieved a substantial benefit from palliative radiotherapy and have not redeveloped symptoms by 12 months post treatment

DETAILED DESCRIPTION:
One third of patients treated in the radiation oncology department are treated with palliative intent. These patients are usually unwell due to their advanced disease and suffering from pain and other symptoms related to bony and soft tissue metastases. Radiation therapy (RT) has an important role in the symptomatic relief and improvement in the quality of life (QoL) for these patients. A meta-analysis of 29 randomised controlled trials (RCTs) estimated the overall response rate (ORR) following RT for bone metastases at approximately 60% with up to one quarter of patients experiencing a complete response (CR). However, palliative patients form a diverse group of patients and selecting the optimal number of palliative treatments which provides an enduring benefit while not being burdensome for the patient can be challenging. The ideal treatment is one that provides lasting symptom control and involves the least number of treatments. Up to one quarter of patients with advanced cancer who undergo palliative RT will die within 1 month of the treatment, while up to 50% of palliative patients will be alive at 12 months . In patients who receive a single fraction of 8Gy, up to 20% of these patients require retreatment to the same site, compared with 8% who receive multiple fraction treatment . One potential option to increase the duration of local control is with hypofractionated, dose escalated radiation.A phase II non-inferiority study investigated this hypothesis in non-spine bone metastases, comparing a single treatment of 12Gy to 30Gy in 10 fractions. The cohort reported a higher pain response in the single fraction dose escalated arm as early as 2 weeks post treatment (62 vs 32%), which was maintained at 9 months (77% vs 46% respectively).

ELIGIBILITY:
Inclusion Criteria:

* Metastatic cancer
* Recommended for 5-10 fractions palliative radiation
* Patients with spinal cord compression are eligible for enrolment

Exclusion Criteria:

* Unwilling or unable to give informed consent
* Patients who are recommended for single fraction palliative radiation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-05-31 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
benefit from palliative radiotherapy | 9 months
  to determine the percentage of patients who have achieved a substantial benefit from palliative radiotherapy and have not redeveloped symptoms by 9 months post treatment

SECONDARY OUTCOMES:
Feasibility of the trial | 2 years
  This will be assessed by the treatment wait time, the amount of time spent in the Radiation Department, the completion rates of electronic Patient Reported Outcome (ePRO)'s and comparing patient and carer assessments
Trial Safety | 2 years
  this will be determined by the radiation dose delivered to organs at risk and patient and carer reported toxicity from treatment
Efficacy of treatment | 2 years
  Efficacy will be determined by reported treatment benefit, pain response, symptom control,re-treatment rates, overall survival and patient and carer regret

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Eade, Principal Investigator — Northern Sydney Cancer Centre, Royal North Shore Hospital
Locations (1):
- Royal North Shore Hospital, Saint Leonards, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: Undecided
The results of this trial will be published in a peer reviewed journal.